CLINICAL TRIAL: NCT04571840
Title: A Study Comparing Bi-parametric MRI to Multi-parametric MRI in the Diagnosis of Clinically Significant Prostate Cancer
Brief Title: Prostate Imaging Using MRI +/- Contrast Enhancement
Acronym: PRIME
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 135819
Record Dates: First submitted 2020-09-09; First posted 2020-10-01 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Prostate Cancer
Keywords: mri; biopsy; targeted; diagnosis; multiparametric; biparametric
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Intervention Model Description: Within-person controlled, paired cohort, diagnostic evaluation study. Participants undergo two index tests and a reference test.
Who Masked: Care Provider
Masking Description: Radiologist assessing MRI for suspicion of prostate cancer is blinded to the contrast sequence when reporting the biparametric MRI. After this report, they are unblinded to the contrast sequence and report the multiparametric MRI. All biopsies conducted as a result of MRI findings will be labelled as bpMRI and mpMRI, and diagnostic accuracy will be assessed against histology findings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- mpMRI (Active Comparator): Multiparametric MRI
  Interventions: Diagnostic Test: Multiparametric MRI +/- prostate biopsy
- bpMRI (Experimental): Biparametric MRI
  Interventions: Diagnostic Test: Biparametric MRI +/- prostate biopsy

INTERVENTIONS:
Diagnostic Test: Multiparametric MRI +/- prostate biopsy — MRI with T2-weighted, diffusion weighted and dynamic contrast enhanced sequences followed by prostate biopsy if indicated on MRI and clinical findings
  Arms: mpMRI
Diagnostic Test: Biparametric MRI +/- prostate biopsy — MRI with T2-weighted and diffusion weighted sequences followed by prostate biopsy if indicated on MRI and clinical findings
  Arms: bpMRI

SUMMARY:
This prospective clinical trial (PRostate Imaging using Mri +/- contrast Enhancement (PRIME)) aims to assess whether biparametric MRI (bpMRI) is non-inferior to multiparametric mpMRI (mpMRI) in the detection of clinically significant prostate cancer.

This means that we are comparing MRI scans that requires injection of IV contrast (the current standard practice) versus MRI scans that can be performed without IV contrast in the detection of prostate cancer.

DETAILED DESCRIPTION:
The PRECISION study (NCT02380027) has established that multiparametric MRI +/- targeted biopsy of suspicious areas identified on MRI is superior to standard 12 core TRUS biopsy in the detection of clinically significant prostate cancer (Gleason > 3+ 4) (38% vs 26%), in reducing the detection of clinically insignificant prostate cancer (Gleason 3 + 3) (9% vs 22%) and in maximising the proportion of cores positive for prostate cancer (44% vs 19%).

Multiparametric MRI (mpMRI) typically uses T2-weighted (T2W), diffusion-weighted (DWI) and dynamic contrast enhanced (DCE) sequences. As a mpMRI is a precious resource, due to capacity and resource limitations, one of the major challenges across institutions is delivering a health service with pre-biopsy MRI before a biopsy in all men with suspected prostate cancer.

However, biparametric MRI (bpMRI), that is, a combination of T2W and DWI, which does not use the DCE sequences, has demonstrated similar detection rates of prostate cancer as mpMRI in some studies and there is a debate about the necessity of the DCE sequence.

The potential advantages of avoiding the DCE sequence include avoiding the cost associated with it, shorter scan time, avoiding the need for medical practitioner attendance, and avoiding putative basal ganglia accumulation and the possibility of adverse neurological effect. Thus, a bpMRI approach may be more feasible and have health-economic benefits over a mpMRI approach and may thus increase the accessibility of this resource to men who need it.

PRIME is a multi-centre study. Men referred with clinical suspicion of prostate cancer based on raised prostate specific antigen (PSA) or abnormal digital rectal examination (DRE) who have had no prior biopsy undergo mpMRI. The DCE sequence is blinded from the radiologist who reports the bpMRI first. After reporting the bpMRI, the DCE sequence is made available to the radiologist who reports the mpMRI. The MRIs and lesions are scored on 1-5 scales of suspicion for the likelihood that clinically significant cancer is present:

1. - Very low (clinically significant cancer is highly unlikely to be present)
2. - Low (clinically significant cancer is unlikely to be present)
3. - Intermediate (the presence of clinically significant cancer is equivocal)
4. - High (clinically significant cancer is likely to be present)
5. - Very high (clinically significant cancer is highly likely to be present)

Men with non-suspicious MRI on bpMRI and mpMRI and low clinical risk of prostate cancer will be counselled by their clinical teams as per routine clinical care. In routine clinical practice these men typically do not undergo prostate biopsy.

Suspicious areas scoring 3, 4 or 5 on either bpMRI or mpMRI will undergo targeted and systematic biopsy using the information from the mpMRI to influence biopsy conduct. Suspicious areas will be labelled by their MRI score, with their location according to sector diagrams.

The proportion of patients with clinically significant prostate cancer will be ascertained and compared between bpMRI and mpMRI.

Treatment eligibility decisions without the DCE information will be made and once the clinicians are unblinded to the DCE sequence the impact that this information makes on the treatment decision will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Men at least 18 years of age referred with clinical suspicion of prostate cancer
2. Serum PSA ≤ 20ng/ml
3. Fit to undergo all procedures listed in protocol
4. Able to provide written informed consent

Exclusion Criteria:

1. Prior prostate biopsy
2. Prior treatment for prostate cancer
3. Prior prostate MRI on a previous encounter
4. Contraindication to MRI
5. Contraindication to prostate biopsy
6. Unfit to undergo any procedures listed in protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of men with clinically significant cancer | When biopsy results available, at an expected average of 30 days post-biopsy

SECONDARY OUTCOMES:
Proportion of men with clinically insignificant cancer (Gleason grade 3+3 / Gleason grade group 1) | When biopsy results available, at an expected average of 30 days post-biopsy
Agreement between bpMRI and mpMRI for score of suspicion | When MRI results available, at an expected average of 30 days post-MRI
  Score of suspicion on MRI (1-5) - lowest score = 1 = highly unlikely to be significant cancer. Highest score = 5 = highly likely to be significant cancer. For MRI to be non-suspicious it needs to be scored 1 or 2 on both Likert and PIRADSv2.1 systems. For MRI to be suspicious it can to be scored 3, 4 or 5 on either Likert or PIRADSv2.1 systems.
Agreement between bpMRI and mpMRI for radiological staging decision | When MRI results available, at an expected average of 30 days post-MRI
Agreement between bpMRI and mpMRI for treatment eligibility | When treatment options discussed in multidisciplinary meeting, at an expected average of 30 days post intervention
  At the coordinating centre, in a multi-disciplinary team meeting, treatment eligibility decisions without the DCE information will be made and once the clinicians are unblinded to the DCE sequence the impact that this information makes on the treatment decision will be evaluated.
Test performance characteristics for bpMRI & mpMRI when using the Likert scoring system in comparison to the PIRADS scoring system | When biopsy results available, at an expected average of 30 days post-MRI
Proportion of men with cancer missed by bpMRI and mpMRI-targeted biopsies and detected by systematic biopsy | When biopsy results available, at an expected average of 30 days post-biopsy
Cost-effectiveness of BpMRI compared to mpMRI (cost per diagnosis of prostate cancer) | At an expected average of 30 days post-intervention
  A within-trial analysis will be conducted to calculate the total cost for bpMRI and mpMRI and mean cost per patient if a strategy of bpMRI or mpMRI were adopted. The cost per diagnosis of clinically significant cancer will be calculated for bpMRI and mpMRI. An incremental cost effectiveness ratio may be calculated by deriving the additional cost per case of clinically significant cancer diagnosed. The cost of avoiding each additional case of clinically insignificant cancer diagnosed may also be calculated. Consideration will be given to extending this analysis using economic modelling to allow a lifetime perspective to be taken and the estimation of quality adjusted life years (QALYs). Costs of procedures will be estimated by multiplying standard unit costs by key resource using data captured within the trial. If possible, standard unit costs (e.g. NHS Reference costs) will be supplemented by unit cost data (and uncertainty around these costs) from the participating trial sites.

CONTACTS AND LOCATIONS:
Overall Officials: Veeru Kasivisvanathan, MBBS PhD, Study Chair — University College, London; Caroline Moore, MD FRCS, Principal Investigator — University College, London; Mark Emberton, MD FRCS, Principal Investigator — University College, London; Clare Allen, FRCR, Principal Investigator — University College London Hospital; Shonit Punwani, PhD FRCR, Principal Investigator — University College, London; Francesco Giganti, MD, Principal Investigator — University College, London
Locations (31):
- United States (4):
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone, New York, New York
  - Icahn School of Medicine (Mount Sinai), New York, New York
  - New York Presbyterian Hospital, New York, New York
- Centro de Urologia, Buenos Aires, Argentina
- Australia (2):
  - Monash University, Melbourne
  - Peter MacCallum Cancer Centre, Melbourne E.
- Ghent University Hospital, Ghent, Belgium
- Hospital Sírio-Libanês, São Paulo, Brazil
- Princess Margaret Cancer Centre, Toronto, Canada
- Herlev and Gentofte Hospital, Copenhagen, Denmark
- Helsinki University Hospital, Helsinki, Finland
- France (3):
  - Bordeaux Pellegrin University Hospital, Bordeaux
  - CHU Lille, Lille
  - Sorbonne Université, Paris
- Germany (4):
  - Heinrich Heine University Düsseldorf, Düsseldorf
  - Essen University Hospital, Essen
  - University Hospital Frankfurt, Frankfurt
  - Martini Klinik, Hamburg
- Italy (4):
  - San Raffaele Hospital, Milan
  - Sapienza University, Rome
  - San Giovanni Battista Hospital, Turin
  - University Hospital of Udine, Udine
- Radboudumc, Nijmegen, Netherlands
- Tan Tock Seng Hospital, Novena, Singapore
- Spain (2):
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario La Moraleja, Madrid
- United Kingdom (4):
  - Addenbrooke's Hospital, Cambridge
  - Royal Free London NHS Foundation Trust, London
  - University College London and University College London Hospital, London
  - Whittington Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be available at request for bona fide researchers with important research questions subject to approval by the study steering committee.
Supporting Information: Study Protocol, SAP
Time Frame: Data will become available 1 year after publication of the main study results.
Access Criteria: A study steering committee will review all requests for access to the data and will make decisions on whether or not to grant access to bona fide researchers based on the importance of the research question being asked, ensuring analysis is non overlapping with existing analyses and planned analyses.

REFERENCES:
- [Derived] Ng ABCD, Asif A, Agarwal R, Panebianco V, Girometti R, Ghai S, Gomez-Gomez E, Budaus L, Barrett T, Radtke JP, Kesch C, De Cobelli F, Pham T, Taneja SS, Hu JC, Tewari A, Rodriguez Cabello MA, Dias AB, Mynderse LA, Borghi M, Boesen L, Singh P, Renard-Penna R, Leow JJ, Falkenbach F, Pecoraro M, Giannarini G, Perlis N, Lopez-Ruiz D, Kastner C, Schimmoller L, Rossiter M, Nathan A, Khetrapal P, Chan VW, Haider A, Clarke CS, Punwani S, Brew-Graves C, Dickinson L, Mitra A, Brembilla G, Margolis DJA, Takwoingi Y, Emberton M, Allen C, Giganti F, Moore CM, Kasivisvanathan V; PRIME Study Group Collaborators. Biparametric vs Multiparametric MRI for Prostate Cancer Diagnosis: The PRIME Diagnostic Clinical Trial. JAMA. 2025 Oct 7;334(13):1170-1179. doi: 10.1001/jama.2025.13722. PMID 40928788
- [Derived] Giganti F, Ng A, Asif A, Chan VW, Rossiter M, Nathan A, Khetrapal P, Dickinson L, Punwani S, Brew-Graves C, Freeman A, Emberton M, Moore CM, Allen C, Kasivisvanathan V; PRIME Quality Improvement Group. Global Variation in Magnetic Resonance Imaging Quality of the Prostate. Radiology. 2023 Oct;309(1):e231130. doi: 10.1148/radiol.231130. PMID 37815448
- [Derived] Asif A, Nathan A, Ng A, Khetrapal P, Chan VW, Giganti F, Allen C, Freeman A, Punwani S, Lorgelly P, Clarke CS, Brew-Graves C, Muirhead N, Emberton M, Agarwal R, Takwoingi Y, Deeks JJ, Moore CM, Kasivisvanathan V; PRIME Trial Group. Comparing biparametric to multiparametric MRI in the diagnosis of clinically significant prostate cancer in biopsy-naive men (PRIME): a prospective, international, multicentre, non-inferiority within-patient, diagnostic yield trial protocol. BMJ Open. 2023 Apr 5;13(4):e070280. doi: 10.1136/bmjopen-2022-070280. PMID 37019486
- [Derived] Ng A, Khetrapal P, Kasivisvanathan V. Is It PRIME Time for Biparametric Magnetic Resonance Imaging in Prostate Cancer Diagnosis? Eur Urol. 2022 Jul;82(1):1-2. doi: 10.1016/j.eururo.2022.02.021. Epub 2022 Mar 8. PMID 35277288